CLINICAL TRIAL: NCT03558685
Title: Weight Loss Diet in the Treatment of Obese Patients With the Metabolic Syndrome
Brief Title: Weight Loss Diet in Obesity With Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0564-08
Record Dates: First submitted 2018-05-31; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Obesity; Diet Modification
MeSH Terms: conditions — Obesity | interventions — Diet, Reducing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diet (Experimental): Nutritional recommendation consisted of moderate caloric restriction, set at 25% to 30% less than calories needed for resting metabolic rate. We applied a high protein Mediterranean diet with the following food group distribution: 30% as protein (> 0.8 g/kg/d); 40% as carbohydrates with medium/low glycemic index; 30% as fat (≥10%monounsaturated fatty acid, ≤7% saturated fatty acid, no trans fats, and 1.6 g omega-3 for men and 1.1 g omega-3 for women). Diet was rich in olive oil, fish, chicken, nuts, white milk products, fruits, and vegetables but low in artificial sugars, commercial sweets, pastries, butter, margarine, and red meat. Dietary fiber content ≥25 g/day
  Interventions: Behavioral: Weight loss diet

INTERVENTIONS:
Behavioral: Weight loss diet — Nutritional recommendation consisted of moderate caloric restriction, set at 25% to 30% less than calories needed for resting metabolic rate. We applied a high protein Mediterranean diet with the following food group distribution: 30% as protein (> 0.8 g/kg/d); 40% as carbohydrates with medium/low glycemic index; 30% as fat (≥10% monounsaturated fatty acid, ≤7% saturated fatty acid, no trans fats, and 1.6 g omega-3 for men and 1.1 g omega-3 for women). Diet was rich in olive oil, fish, chicken, nuts, white milk products, fruits, and vegetables but low in artificial sugars, commercial sweets, pastries, butter, margarine, and red meat. Dietary fiber content ≥25 g/day

SUMMARY:
Concomitant interventions included lifestyle modification with a personally tailored program of diet as detailed below and physical activity adjusted for age and specific physical limitations, targeting engagement in physical activity of at least 150 minutes/week. Lipid lowering and or blood pressure lowering drugs were prescribed as needed according to guideline-assisted medical practice. Patients were seen by a physician every 3 month. The dietitian had a weekly meeting with the patients for the first three months, every other week during months 4-6, once a month during month 7-9 and every 6 weeks during the last three months of the study.

ELIGIBILITY:
Inclusion Criteria:

- fulfilled the diagnostic criteria for the metabolic syndrome as defined by the Third Report of the Adult Treatment Panel (ATPIII).

Exclusion Criteria:

* diabetes
* the presence of current or recent pregnancy or intention to conceive within the trial's period
* chronic renal or liver disease
* past bariatric surgery
* current participation in any dietary/ medical program with current continuous weight loss.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
% BMI Change | One Year, from the initiation of the intervention to its termination.
  BMI is calculated as weight in Kg divided by height in meters X height in meters. Percent change will be calculated as the difference in BMI units (kg/m2) between the final BMI and the initial BMI, divided by the initial BMI, multiplied by 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Naftali Stern, MD, Principal Investigator — Institute of Endocrinology, Metabolism and Hypertension Tel Aviv-Sourasky Medical Center